CLINICAL TRIAL: NCT00119613
Title: A Randomized, Double Blind, Placebo-Controlled Study of Subjects With Previously Untreated Extensive-Stage Small-Cell Lung Cancer (SCLC) Treated With Platinum Plus Etoposide Chemotherapy With or Without Darbepoetin Alfa
Brief Title: A Study of Subjects With Previously Untreated Extensive-Stage Small-Cell Lung Cancer (SCLC) Treated With Platinum Plus Etoposide Chemotherapy With or Without Darbepoetin Alfa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20010145
Record Dates: First submitted 2005-07-07; First posted 2005-07-14 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Small Cell Lung Cancer
Keywords: Oncology; Clinical Trial; Hemoglobin; Darbepoetin alfa; Survival; Carboplatin; Cisplatin; Etoposide; Extensive Stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group 1 - darbepoetin alfa (Experimental): Darbepoetin alfa 300 mcg QW for the first 4 weeks, followed by Q3W dosing commencing on week 5 for the remainder of the treatment period.
  Interventions: Drug: darbepoetin alfa
- Group 2 - Placebo (Placebo Comparator): Placebo QW for the first 4 weeks, followed by Q3W dosing commencing on week 5 for the remainder of the treatment period.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — placebo
  Arms: Group 2 - Placebo
Drug: darbepoetin alfa — darbepoetin alfa
  Arms: Group 1 - darbepoetin alfa

SUMMARY:
The purpose of this study is to evaluate whether increasing or maintaining hemoglobin concentrations with darbepoetin alfa, when administered with platinum-containing chemotherapy in subjects with previously untreated extensive-stage small cell lung cancer (SCLC), increases survival.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven SCLC, extensive-stage
* Planned to receive chemotherapy of carboplatin or cisplatin plus etoposide every 3 weeks for 6 cycles
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Life expectancy greater than or equal to 3 months
* Hemoglobin concentration greater than or equal to 9.0 g/dL and less than or equal to 13g/dL
* Adequate renal, liver and hematopoietic function
* Subjects must sign and date a written Institutional Review Board /Independent Ethics Committee-approved Informed Consent Form

Exclusion Criteria:

* Known primary hematologic disorder which could cause anemia
* Brain metastases that are either symptomatic or treated with medications
* Unstable or uncontrolled disease/condition, related to or affecting cardiac function
* Other known primary malignancy within the past 5 years with the exception of curatively treated basal cell carcinoma, squamous cell carcinoma in situ cervical carcinoma or surgically cured malignancies
* Iron deficiency
* Known positive test for human immunodeficiency virus infection
* Received greater than 2 units of packed red blood cells within 4 weeks of randomization or any RBC transfusions within 2 weeks before randomization
* Received rHuEPO or darbepoetin alfa therapy within 4 weeks of randomization
* Previous chemotherapy for SCLC
* Previous radiotherapy except as symptom palliation for bone or brain lesions and at least 24 hours since prior radiotherapy for symptom palliation providing extent of radiotherapy makes marked bone marrow suppression unlikely
* Less than 30 days since receipt of any drug or device that is not approved for any indication
* Pregnant or breast-feeding
* Not using adequate contraceptive precautions
* Previously randomized into this study
* Known hypersensitivity to recombinant mammalian-derived product or any other ingredients contained in the study drug
* Any medical, mental, or other conditions that makes the subject unsuitable for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2002-12; Primary Completion 2007-01 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin concentration from baseline to the end of the chemotherapy treatment period | from baseline to the end of the chemotherapy treatment period
Survival time

SECONDARY OUTCOMES:
Change in FACT-fatigue subscale scores from baseline to the end of study treatment | from baseline to the end of study treatment
Incidence of Adverse Events (including serious and treatment related) | Throughout study
Changes in laboratory values, changes in vital signs and incidence of concomitant medications | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Pirker R, Ramlau RA, Schuette W, Zatloukal P, Ferreira I, Lillie T, Vansteenkiste JF. Safety and efficacy of darbepoetin alpha in previously untreated extensive-stage small-cell lung cancer treated with platinum plus etoposide. J Clin Oncol. 2008 May 10;26(14):2342-9. doi: 10.1200/JCO.2007.15.0748. PMID 18467726
- [Derived] Ventz S, Khozin S, Louv B, Sands J, Wen PY, Rahman R, Comment L, Alexander BM, Trippa L. The design and evaluation of hybrid controlled trials that leverage external data and randomization. Nat Commun. 2022 Oct 2;13(1):5783. doi: 10.1038/s41467-022-33192-1. PMID 36184621
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20010145_Clinical_Trial_Posting.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20010145_Clinical_Trial_Posting_Apr_20.pdf